CLINICAL TRIAL: NCT04728113
Title: Early Integration of Supportive Care Into Standard Oncology Care for Metastatic Uveal Melanoma Patients
Brief Title: Early Integration of Supportive Care for Metastatic Uveal Melanoma Patients (EarlyTogether)
Acronym: EARLY TOGETHER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IC 2019-09
Record Dates: First submitted 2021-01-08; First posted 2021-01-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-02

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early together group (Experimental): Oncological standard of care at M0, M3, M6, M9 and M12 with early introduction of supportive care every 6 weeks.
  Interventions: Other: Supportive care visit with questionnaires; Other: Oncological standard visit
- Control group (Active Comparator): Oncological standard of care at M0, M3, M6, M9 and M12.
  Interventions: Other: Oncological standard visit

INTERVENTIONS:
Other: Supportive care visit with questionnaires — 5 Questionnaires (SCNS, QLQ-C30, HADS, PTPQ, GSE) will be filled by the patient with introduction of supportive care visit
  Arms: Early together group
Other: Oncological standard visit — Oncological standard visit

SUMMARY:
The study main objective is to assess whether the early introduction of supportive care demonstrates a benefit on patients' psychological care needs at 6 months (M6), versus oncological standard of care in patients with metastatic UM.

Supportive care in patients with metastatic Uveal Melanoma (UM)

DETAILED DESCRIPTION:
Before the start of the study, medical oncologists and supportive care physicians from both the sites will attend Communication Skills Training (CST) workshops provided by an expert team in the field. The training sessions will focus on practicing the required communication skills needed in consultations.

The randomization will assign patients, with a 1:2 ratio, to "Introduction of supportive care when medically needed" (Arm A: Control Group) or "Initial concomitant management by the oncologist and the supportive care team" (Arm B: Early Together Group).

Selected and validated questionnaires will be filled at baseline, 6 and 12 months by the patients before the consultation, in the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients with metastatic UM;
2. no surgery or loco-regional treatment of metastases in a curative intent;
3. systemic treatment planned or started since less than 2 months;
4. ECOG PS 0-1;
5. no uncontrolled symptoms;
6. liver function tests in normal range or ≤ grade 2;
7. signed informed consent;
8. able to fill the questionnaires.

Exclusion Criteria:

1. patient<18 years old;
2. patient condition requiring supportive care before any systemic specific treatment for metastases;
3. acute psychopathological disorder incompatible with the study;
4. prior medical condition incompatible with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-01-22 (Actual)

PRIMARY OUTCOMES:
34 items - Supportive Care Needs Survey | 6 months
  The main study criterion is the score to the "Care and Support Needs" domain (items 18-22) of the SCNS-SF34 questionnaire obtained in the two arms at 6 months after inclusion. A 10 points mean score difference expected between groups. Each question is ranged from 0 (no need of supportive care) to 5 (strong need of supportive care). Scores for Outcome 1 may vary from 0 to 25.

CONTACTS AND LOCATIONS:
Overall Officials: PIPERNO NEUMAN Sophie, MD, Principal Investigator — Institut Curie
Locations (2):
- France (2):
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).